CLINICAL TRIAL: NCT02311816
Title: Increase in Procalcitonin Kinetics May be a Good Indicator of Starting Empirical Antibiotic Treatment in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Domonkos Trásy (Other)
Responsible Party: Sponsor-Investigator, Domonkos Trásy, Ph.D. student; Department of Anaesthesiology and Intensive Therapy, Szeged University
Organization: Szeged University (Other)
Other Study IDs: PCT-infection
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Bacterial Infection
Keywords: Bacterial infection, empiric antibiotic therapy
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infection: Based on the microbiological results and clinical picture patients were grouped post hoc into "infection" and "no infection" groups by two independent experts (intensivist, infectologist) who were blinded for procalcitonin.
- No infection: Based on the microbiological results and clinical picture patients were grouped post hoc into "infection" and "no infection" groups by two independent experts (intensivist, infectologist) who were blinded for procalcitonin.

SUMMARY:
The value of procalcitonin change from the day before to the day when infection was suspected in predicting bacterial infection in intensive care patients.

DETAILED DESCRIPTION:
Starting antibiotic therapy early in critically ill patients with suspected infection is of utmost importance with significant effect on survival. Procalcitonin is a reliable sepsis marker but results about its usefulness in initiating antimicrobials are conflicting. Our aim is to investigate the predictive value of 24 hours procalcitonin kinetics before starting empirical antibiotic therapy in intensive care patients as an indicator of the presence of bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of infection
* Suspected or proven acute infection requiring empiric antibiotic therapy as decided by the attending ICU physician
* Microbiological sample sent for staining
* Inflammatory markers available from the previous day

Exclusion Criteria:

* Patients younger than 18 years
* Who received prophylactic or empiric antibiotic therapy 48 hours before inclusion
* Whose receiving acute renal replacement therapy in the first 24 hours following antibiotic treatment
* Following cardiopulmonary resuscitation
* End stage diseases with a "do not resuscitate" order
* Immunocompromised patients (human immunodeficiency virus infection, bone marrow transplantation, malignant haematological disorders and chemotherapy)
* Post cardiac surgery patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspected infection during their stay on the intensive care unit were screened for eligibility. Patients were enrolled, when the attending intensive care specialist had a suspicion of infection and decided to start empirical antibiotic therapy and infalmmatory markers were available from the previous day.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2012-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Procalcitonin kinetic | 24 hours before starting empiric antibiotic treatment
  Procalcitonin levels are measured at starting empiric antibiotic treatment and 24 hours before. The changes in percentage are calculated form the day before and right before the first exposition of the antibiotic therapy.

SECONDARY OUTCOMES:
C-reactive protein kinetic | 24 hours before starting empiric antibiotic treatment
  C-reactive protein levels are measured at starting empiric antibiotic treatment and 24 hours before. The changes in percentage are calculated form the day before and right before the first exposition of the antibiotic therapy.
Body temperature kinetic | 24 hours before starting empiric antibiotic treatment
  Body temperatures are measured at starting empiric antibiotic treatment and 24 hours before. The changes in percentage are calculated form the day before and right before the first exposition of the antibiotic therapy.
White blood cell count kinetic | 24 hours before starting empiric antibiotic treatment
  White blood cell count levels are measured at starting empiric antibiotic treatment and 24 hours before. The changes in percentage are calculated form the day before and right before the first exposition of the antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Therapy, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Derived] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z. Delta Procalcitonin Is a Better Indicator of Infection Than Absolute Procalcitonin Values in Critically Ill Patients: A Prospective Observational Study. J Immunol Res. 2016;2016:3530752. doi: 10.1155/2016/3530752. Epub 2016 Aug 15. PMID 27597981